CLINICAL TRIAL: NCT00844493
Title: Validation of Low-dose ETEC Challenge Model in U.S. Adults and Re-challenge of Immune Subjects With a Homologous ETEC Strain (H10407)
Brief Title: Low-dose Challenge Model With Enterotoxigenic E Coli
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: PATH Vaccine Solutions (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CIR259
Record Dates: First submitted 2009-02-13; First posted 2009-02-16 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2013-04

CONDITIONS: Diarrhea
Keywords: diarrhea; vaccine; enterotoxigenic E coli; colonization factor antigen; volunteer study
MeSH Terms: conditions — Diarrhea | interventions — Buffers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- H10407 challenge 1 (Experimental): 7 or 8 logs of E. coli strain H10407 with CeraVacx buffer
  Interventions: Biological: E coli strain H10407 and buffer
- H10407 challenge 2 (Experimental): 7 or 8 logs of E. coli strain H10407 with bicarbonate buffer
  Interventions: Biological: E coli strain H10407 and buffer
- H10407 challenge 3 (Experimental): 6 logs of E. coli H10407 with bicarbonate buffer
  Interventions: Biological: E coli strain H10407 and buffer
- H10407 challenge 4 (Experimental): 5 logs of E. coli H10407 with bicarbonate buffer
  Interventions: Biological: E coli H10407 and buffer

INTERVENTIONS:
Biological: E coli strain H10407 and buffer — 7 or 8 logs of the bacteria with bicarbonate buffer
  Arms: H10407 challenge 1
Biological: E coli strain H10407 and buffer — Bacteria in a dose of 8 logs with CeraVacx buffer
  Arms: H10407 challenge 2
Biological: E coli strain H10407 and buffer — Bacteria in a dose of 7 logs and CeraVacx buffer
  Arms: H10407 challenge 3
Biological: E coli H10407 and buffer — Bacteria in a dose of 8 logs with bicarbonate buffer
  Arms: H10407 challenge 4

SUMMARY:
This study will validate a model for testing new vaccines designed to protect against intestinal infections with enterotoxigenic Escherichia coli (ETEC). ETEC is one of the most common causes of diarrhea in developing countries and is a common cause of travelers diarrhea. Vaccines are now being developed and their development will be facilitated if we have a valid model for testing these vaccines in human volunteers. We anticipate that the new vaccines will be given to volunteers and they will then be given a dose of virulent ETEC bacteria. If the vaccine is effective, the volunteers should not development diarrhea, but if the vaccine is not effective, the volunteers will have diarrhea for a few days.

During this study, we will validate a minimum dose of virulent ETEC bacteria which is sufficient to cause diarrhea in healthy adult volunteers and to identify conditions that can make this model reliable.

We will also determine, in a follow-up group of volunteers, if being exposed to the ETEC bacteria previously will protect against a subsequent illness when they are exposed to the same bacteria a second time. We believe that the previously exposed group will be protected and we will study the immune response to these exposures to help design vaccines that can accomplish this kind of protection.

DETAILED DESCRIPTION:
This is a study in which healthy adult inpatient volunteers will be challenged with Escherichia coli, strain H10407 using different conditions. The study has the following objectives.

1. To identify a revised set of procedures for the ETEC H10407 challenge model that will allow for an inoculum dose <108 organisms, and that will cause diarrhea in 50% or more of subjects without causing high output diarrhea, as determined by stool output volumes or signs and symptoms associated with hypovolemia.
2. To measure mucosal and systemic immune responses to ETEC H10407 in naïve and immune subjects.
3. To determine the extent to which recent enteric illness due to ETEC H10407will protect subjects against diarrhea when re-challenged with H10407.
4. To determine the extent to which mucosal and/or systemic antibody responses following ETEC H10407diarrhea are predictive of protection in a re-challenge study.

The study is divided into 4 cohorts. The first cohort will test four conditions of dose and buffer for the challenge. Using the conditions that appear to be best, a larger number of volunteers will be given this challenge to validate these conditions. The third group will be divided between some volunteers who had been ill during previous studies and some who have not been exposed before.

Specimens will be obtained to determine the extent of excretion of the challenge strain and the immune responses to the challenge. These will include measures of both systemic and local intestinal immunity.

Update as of May 2010:

The clinical portion of the study has been completed and is no longer recruiting. The overall results were presented at two meetings including the Vaccines for Enteric Diseases in Spain in 2009 and the US-Japan Medical Science conference on Cholera and Enteric Disease in San Diego in 2009. Volunteers who received the lower dose (7 logs), along with an overnight fast developed diarrhea with an attack rate of >75%. Volunteers who were challenged a second time with this dose were protected from subsequent illness. Immunological assessment of the volunteers is continuing.

Update as of November 2011 Results of the first three cohorts were published in 2011 (see citation below). A fourth cohort is planned to be enrolled to evaluate the virulence of an even lower dose of 5 and 6 logs of E coli. The same procedures will be carried out as with earlier cohorts.

Update as of April 2013 Following challenge with 5 or 6 logs of strain H10407, the attack rates were lower (approximately 30%). Among those volunteers who did develop illness, the severity was the same as with higher doses. completion of these lower doses completes the dose response curve for H10407. For future challenge studies, 7 logs of H10407 with bicarbonate buffer will be used.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between 18 and 45 years of age, inclusive.
2. General good health, as determined by physical exam, laboratory testing, and medical history.
3. Laboratory values within acceptable range for complete blood count (CBC), Alanine Aminotransferase (ALT), and serum creatinine as determined by PI.
4. Demonstrate comprehension of the protocol procedures and knowledge of ETEC illness by passing a written examination (pass grade ≥ 70%)
5. Able and willing to sign an informed consent.
6. Available to participate for the length of the study.
7. Female only: Females of childbearing potential will use an effective method of contraception during the study, including abstinence, hormonal contraception, barrier, implantables or injectables.

Exclusion Criteria:

1. Presence of a clinically significant medical condition (including but not limited to any chronic illnesses, immunosuppressive illness, cancer, diabetes, gastrointestinal disease, such as peptic ulcer, symptoms or evidence of active gastritis or gastroesophageal reflux disease, inflammatory bowel disease)
2. Evidence of immunoglobulin A (IgA) deficiency (serum IgA <5 or limit of detection of assay)
3. Evidence of HIV, hepatitis B virus (HBV), hepatitis C virus (HCV), by medical history or laboratory testing.
4. Symptoms consistent with Traveler's Diarrhea concurrent with travel to countries where ETEC or cholera infection is endemic (most of the developing world) within two years prior to receipt of investigational agent, OR planned travel to endemic countries during the length of the trial.
5. History of significant psychiatric illness requiring hospitalization or any suicide attempts within the past 2 years.
6. History of significant drug or alcohol abuse requiring hospitalization or rehabilitation within the past 2 years.
7. Evidence of significant drug abuse, as determined by the Principal Investigator, on toxicity screening.
8. Fewer than 3 stools per week or more than 3 stools per day as the usual frequency; loose or liquid stools other than on an occasional basis.
9. History of allergic reaction to fluoroquinolones, cotrimoxazole, or ampicillin/penicillin (excluded if allergic to two of three).
10. History of diarrhea in the 2 weeks prior to receipt of investigational agent.
11. Weekly use of laxatives or any agent that increases gastric pH.
12. Use of antibiotics during the 7 days prior to receipt of investigational agent.
13. Use of proton pump inhibitors, H2 blockers, or antacids within 48 hours of receipt of investigational agent.
14. History of vaccination for or ingestion of ETEC, cholera, or heat labile toxin (LT) toxin within 5 years.*
15. History of participation in prior ETEC H10407 research studies.*
16. Use of any other investigational product within 30 days preceding the receipt of investigational agent, or planned use during the active study period.
17. Use of any medication known to affect the immune function (e.g., corticosteroids) within 30 days preceding receipt of investigational agent or planned use during the active study period. (Topical and intra-articular steroids will not exclude subjects).
18. Any other condition, which in the opinion of the investigator, could affect subject safety or interfere with the trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2009-02; Primary Completion 2012-02 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Occurrence of moderate or severe diarrhea | 5 days

SECONDARY OUTCOMES:
Antibody response to Cholera toxin b subunit, Lipopolysaccharide and colonization factor antigen | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Clayton Harro, M.D., Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Center for Immunization Research, Johns Hopkins Bloomberg School of Public Heatlh, Baltimore, Maryland, United States

REFERENCES:
- [Background] McKenzie R, Bourgeois AL, Engstrom F, Hall E, Chang HS, Gomes JG, Kyle JL, Cassels F, Turner AK, Randall R, Darsley M, Lee C, Bedford P, Shimko J, Sack DA. Comparative safety and immunogenicity of two attenuated enterotoxigenic Escherichia coli vaccine strains in healthy adults. Infect Immun. 2006 Feb;74(2):994-1000. doi: 10.1128/IAI.74.2.994-1000.2006. PMID 16428745
- [Background] Sack DA, Shimko J, Sack RB, Gomes JG, MacLeod K, O'Sullivan D, Spriggs D. Comparison of alternative buffers for use with a new live oral cholera vaccine, Peru-15, in outpatient volunteers. Infect Immun. 1997 Jun;65(6):2107-11. doi: 10.1128/iai.65.6.2107-2111.1997. PMID 9169739
- [Background] DuPont HL, Formal SB, Hornick RB, Snyder MJ, Libonati JP, Sheahan DG, LaBrec EH, Kalas JP. Pathogenesis of Escherichia coli diarrhea. N Engl J Med. 1971 Jul 1;285(1):1-9. doi: 10.1056/NEJM197107012850101. No abstract available. PMID 4996788
- [Background] Qadri F, Saha A, Ahmed T, Al Tarique A, Begum YA, Svennerholm AM. Disease burden due to enterotoxigenic Escherichia coli in the first 2 years of life in an urban community in Bangladesh. Infect Immun. 2007 Aug;75(8):3961-8. doi: 10.1128/IAI.00459-07. Epub 2007 Jun 4. PMID 17548483
- [Background] Qadri F, Ahmed T, Ahmed F, Begum YA, Sack DA, Svennerholm AM; PTE Study Group. Reduced doses of oral killed enterotoxigenic Escherichia coli plus cholera toxin B subunit vaccine is safe and immunogenic in Bangladeshi infants 6-17 months of age: dosing studies in different age groups. Vaccine. 2006 Mar 6;24(10):1726-33. doi: 10.1016/j.vaccine.2005.08.110. Epub 2005 Oct 10. PMID 16257098
- [Background] Qadri F, Svennerholm AM, Faruque AS, Sack RB. Enterotoxigenic Escherichia coli in developing countries: epidemiology, microbiology, clinical features, treatment, and prevention. Clin Microbiol Rev. 2005 Jul;18(3):465-83. doi: 10.1128/CMR.18.3.465-483.2005. PMID 16020685
- [Result] Harro C, Chakraborty S, Feller A, DeNearing B, Cage A, Ram M, Lundgren A, Svennerholm AM, Bourgeois AL, Walker RI, Sack DA. Refinement of a human challenge model for evaluation of enterotoxigenic Escherichia coli vaccines. Clin Vaccine Immunol. 2011 Oct;18(10):1719-27. doi: 10.1128/CVI.05194-11. Epub 2011 Aug 18. PMID 21852546
- [Derived] Chakraborty S, Harro C, DeNearing B, Brubaker J, Connor S, Maier N, Dally L, Flores J, Bourgeois AL, Walker R, Sack DA. Impact of lower challenge doses of enterotoxigenic Escherichia coli on clinical outcome, intestinal colonization and immune responses in adult volunteers. PLoS Negl Trop Dis. 2018 Apr 27;12(4):e0006442. doi: 10.1371/journal.pntd.0006442. eCollection 2018 Apr. PMID 29702652
- See also: resource for vaccines for Enterotoxigenic E coli — http://www.path.org/vaccineresources/shigella-etec.php
- See also: web site for the International Centre for Diarrhoeal Disease Research, Bangladesh where much of the work on ETEC is done — http://www.icddrb.org